

# Study Protocol

# The Effect of Milk-Derived Protein Supplementation on the Recovery of Muscle Function following Resistance Exercise

# Project context.

In order to maximise training adaptation during a resistance exercise program effective recovery is critical. Exercise-induced muscle damage (EIMD) occur following resistance exercise and, whilst this can lead to positive training effects e.g. increased muscle size, speed & strength, EIMD may also cause muscle soreness & inflammation that have detrimental effects on training and performance.

#### **Research Question:**

This study aims to analyse the use milk-derived protein supplementation for effective recovery of muscle following resistance exercise.

## **Study Protocol:**

All aspects of the study and risks involved will be explained clearly to all involved.

This study requires **17 DAYS** split into 2 distinct phases, illustrated in Figure 1 and described below. The study will be conducted in the PESS Building at the University of Limerick.



# Phase 1: Days 1 - 8

- I. Food and fluid intake for every eating occasion, every day for days 1 to 7 under the guidance of a qualified dietician/sports nutritionist.
- II. familiarisation resistance exercise / muscle function sessions (around 1 hour each)

Ethical Approval Code: 2016\_12\_09\_EHS

#### Day 1:

Pre-screening: Each subject will undertake preliminary screening consisting of:

- i. medical history and examination by a clinician
- ii. blood sample (SS023) to be evaluated for health-related contraindications
- iii. body composition measurement by DXA to determine whole body and segmental lean tissue mass (SS077);
- iv. exercise training log (6 month recall)
- v. dietary consultation
- vi. habitual physical activity level assessed by EPAQ-2

Day 2 - 8: Subject will be "free-living" during this time. Record of dietary intake under the guidance of a qualified dietitian and sports nutritionist. Physical activity recorded by an exercise physiologist and strength and conditioning coach.

# Phase 2: Days 9 - 17

## Day 9:

- i. Familiarisation sessions to the testing procedures (EHSREC10-RA04, SS014, SS003, SS017, SS035)
- ii. A single blood sample (5ml) will be drawn (SS203).

# Day 10:

I. In the afternoon 200ml of water containing deuterium (heavy water) will be consumed. A small saliva sample will be collected before and 1 hour after consuming the water.

**Days 11-1:** A prescribed diet (gratis) is provided. The meal plan (3 meals, 2 snacks, 1 'shake' per day) based on the habitual dietary intake of resistance-trained athletes and standardised to body mass (Table).

| | Day 1 | Day 2 | Day 3 | Day 4 | Day 5 | Day 6 |
|---|---|---|---|---|---|---|
| Breakfast | Porridge made with<br>water and coconut<br>oil topped with<br>banana and dried<br>cranberries | Scramble eggs with toasts and avocado | Milk & yoghurt<br>shake with fruits,<br>toasts with peanut<br>butter | Porridge made with milk, seeds and nuts | Omelette with<br>mushrooms and<br>vegetables, toasts<br>with butter | Poached eggs, with<br>grilled back bacon,<br>sandwich with<br>vegetables |
| Lunch | Beef burger with<br>multigrain bun and<br>vegetables | Wrap with chicken and vegetables | Chicken curry with brown rice | Roasted pork chops<br>with lettuce salad and<br>mashed potatoes | Beef stir-fry with vegetables and rice | Roasted pork chop<br>with beetroot salad<br>and sweet potatoes<br>wedges |
| Snack | - | Yoghurt with oats<br>and fruits | Sandwich with ham,<br>yoghurt | Pasta with pesto and turkey | Sandwiches with<br>ham cheese and<br>vegetables | Chicken salad with<br>sweet potatoes and<br>sauce based on<br>mayonnaise |
| Dinner | Chicken Breast in<br>the sauce with<br>spinach and potato<br>wedges | Beef stew | Beef steak with<br>green beans and<br>mashed potatoes | Chicken breast with rice, sauce and broccoli | Tuna salad with<br>bread on the side | Spaghetti Bolognese |
| Pre-bed<br>snack | Yoghurt with mixed<br>nuts, honey and<br>pear | Smoothie with protein milk, banana and berries | Cottage cheese, toast<br>with butter and sliced<br>tomatoes | Chocolate milk with a banana | Milk , Weetabix and<br>a mandarin | Yoghurt with<br>crunchy cereal<br>clusters and dried<br>fruits |

# Day 11:

- I. A fasted venous blood sample (5ml; by venepuncture) is drawn and saliva sample collected.
- II. A micro-muscle biopsy sample will be taken from the outside portion of the thigh

Ethical Approval Code: 2016\_12\_09\_EHS

- III. A prescribed protein supplement will be ingested
- IV. A prescribed resistance-exercise Training bout will be completed
- V. 3-hours later a 2<sup>nd</sup> micro-muscle biopsy sample will be taken from the outside portion of the thigh

#### Day 12:

- I. A fasted venous blood sample (5ml; by venepuncture) is drawn and saliva sample collected.
- II. A series of muscle function tests will be conducted
- III. A prescribed protein supplement will be ingested
- IV. No further exercise is permitted

### Day 13:

- V. A fasted venous blood sample (5ml; by venepuncture) is drawn and saliva sample collected.
- VI. A series of muscle function tests will be conducted
- VII. A prescribed resistance-exercise Training bout will be completed
- VIII. A prescribed protein supplement will be ingested
- IX. No further exercise is permitted

# Day 14:

- I. A fasted venous blood sample (5ml; by venepuncture) is drawn and saliva sample collected.
- II. A series of muscle function tests will be conducted
- III. A prescribed protein supplement will be ingested
- IV. No further exercise is permitted

#### Day 15:

- I. A fasted venous blood sample (5ml; by venepuncture) is drawn and saliva sample collected.
- II. A series of muscle function tests will be conducted
- III. A prescribed resistance-exercise Training bout will be completed
- IV. A prescribed protein supplement will be ingested
- V. No further exercise is permitted

# Day 16:

- I. A fasted venous blood sample (5ml; by venepuncture) is drawn and saliva sample collected.
- II. A series of muscle function tests will be conducted
- III. A prescribed protein supplement will be ingested
- IV. No further exercise is permitted

# Day 17:

- I. A fasted venous blood sample (5ml; by venepuncture) is drawn and saliva sample collected.
- II. A series of muscle function tests will be conducted